CLINICAL TRIAL: NCT00389818
Title: A Phase II Trial of Doxil, Rituximab, Cyclophosphamide, Vincristine, and Prednisone (DR-COP) in Patients With Newly Diagnosed AIDS-Associated B-Cell Non-Hodgkin's Lymphoma
Brief Title: Combination Chemotherapy and Rituximab in Treating Patients With Newly Diagnosed AIDS-Related B-Cell Non-Hodgkin's Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AIDS Malignancy Consortium (Network)
Collaborators: National Cancer Institute (NCI) (NIH); The Emmes Company, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AMC-047; U01CA070019 (NIH); CDR0000507634 (Other: NCI)
Record Dates: First submitted 2006-10-18; First posted 2006-10-19 (Estimated); Results first posted 2012-06-29 (Estimated); Last update posted 2018-06-06 (Actual); Status verified 2018-05

CONDITIONS: Lymphoma
Keywords: contiguous stage II grade 3 follicular lymphoma; noncontiguous stage II grade 3 follicular lymphoma; stage I grade 3 follicular lymphoma; stage III grade 3 follicular lymphoma; stage IV grade 3 follicular lymphoma; AIDS-related diffuse large cell lymphoma; contiguous stage II adult diffuse large cell lymphoma; noncontiguous stage II adult diffuse large cell lymphoma; stage I adult diffuse large cell lymphoma; stage III adult diffuse large cell lymphoma; stage IV adult diffuse large cell lymphoma; AIDS-related immunoblastic large cell lymphoma; contiguous stage II adult immunoblastic large cell lymphoma; noncontiguous stage II adult immunoblastic large cell lymphoma; stage I adult immunoblastic large cell lymphoma; stage III adult immunoblastic large cell lymphoma; stage IV adult immunoblastic large cell lymphoma; AIDS-related peripheral/systemic lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Follicular; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Large-Cell, Immunoblastic | interventions — Filgrastim; pegfilgrastim; Rituximab; sargramostim; Cyclophosphamide; Prednisone; Vincristine; Immunohistochemistry

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- DR-COP (Experimental): Single arm interventional study: all subjects receive DR-COP regimen.
  Interventions: Biological: filgrastim; Biological: pegfilgrastim; Biological: rituximab; Biological: sargramostim; Drug: cyclophosphamide; Drug: pegylated liposomal doxorubicin hydrochloride; Drug: prednisone; Drug: vincristine sulfate; Other: immunohistochemistry staining method; Other: laboratory biomarker analysis

INTERVENTIONS:
Biological: filgrastim — Supportive therapy: GF therapy with G-CSF, GM-CSF, or pegfilgrastim will be used in all patients, beginning on Day 3 of each cycle, until post nadir of blood counts from each chemotherapy cycle.
Biological: pegfilgrastim — GF therapy with G-CSF, GM-CSF, or pegfilgrastim will be used in all patients, beginning on Day 3 of each cycle, until post nadir of blood counts from each chemotherapy cycle.
Biological: rituximab — 375 mg/m2 IV Day 1 of each cycle
Biological: sargramostim — GF therapy with G-CSF, GM-CSF, or pegfilgrastim will be used in all patients, beginning on Day 3 of each cycle, until post nadir of blood counts from each chemotherapy cycle.
Drug: cyclophosphamide — 750 mg/m2 IV Day 1 of each cycle
Drug: pegylated liposomal doxorubicin hydrochloride — 40 mg/m2 IV Day 1 of each cycle
Drug: prednisone — 100 mg PO Days 1-5 of each cycle
Drug: vincristine sulfate — 1.4 mg/m2 IV Day 1 (2.0 mg maximum) of each cycle
Other: immunohistochemistry staining method — tissue specimen collected at baseline
Other: laboratory biomarker analysis — tissue specimen collected at baseline

SUMMARY:
RATIONALE: Drugs used in chemotherapy work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Monoclonal antibodies, such as rituximab, can block cancer growth in different ways. Some find cancer cells and help kill them or carry cancer-killing substances to them. Others interfere with the ability of cancer cells to grow and spread. Giving combination chemotherapy together with rituximab may kill more cancer cells.

PURPOSE: This phase II trial is studying how well giving combination chemotherapy together with rituximab works in treating patients with newly diagnosed AIDS-related B-cell non-Hodgkin's lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the complete response rate (complete response and complete response unconfirmed) in patients with newly diagnosed, AIDS-related B-cell non-Hodgkin's lymphoma treated with doxorubicin hydrochloride liposome, rituximab, cyclophosphamide, vincristine, and prednisone (DR-COP).
* Determine the duration of response (relapse-free survival) in patients treated with this regimen.
* Determine the median survival time of patients treated with this regimen.
* Determine rate of bacterial, fungal, and opportunistic infections in patients treated with this regimen.

Secondary

* Determine, preliminarily, the relationship between MDR-1 expression in tumor tissue and response to therapy in patients treated with this regimen.
* Determine, preliminarily, any relationship between response and survival and BCL-2 expression in tumor tissue in patients treated with this regimen.
* Determine any relationship between development of bacterial, fungal, and/or opportunistic infections and baseline CD4 lymphocyte count, HIV-1 RNA level, and quantitative immunoglobulin levels, or changes in quantitative immunoglobulin levels over time in patients treated with this regimen.
* Compare the results of positron emission tomography (PET) scanning with traditional CT scans in predicting response to therapy in these patients.
* Examine the relationship between chemotherapeutic drug levels and receipt of specific antiretroviral and/or anti-infective medications in these patients.
* Examine the mortality and the causes of death in patients treated with this regimen.
* Determine event-free survival at 1 year.

OUTLINE: This is a nonrandomized, multicenter study.

Patients receive doxorubicin hydrochloride liposome IV over 90 minutes, rituximab IV over 5-7 hours, cyclophosphamide IV over 1 hour, and vincristine IV over 1-2 minutes on day 1 and oral prednisone on days 1-5. Patients also receive filgrastim (G-CSF), sargramostim (GM-CSF), or pegfilgrastim beginning on day 3 and continuing until blood counts recover. Treatment repeats every 21-28 days for up to 8 courses in the absence of disease progression or unacceptable toxicity.

Patients undergo laboratory/biomarker studies at baseline and after every 2 courses of chemotherapy. Tissue is examined by immunohistochemistry for BCL-2, Ki67, and MDR-1, along with other markers.

After completion of study treatment, patients are followed periodically for 3 years.

PROJECTED ACCRUAL: A total of 44 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed AIDS-related B-cell non-Hodgkin's lymphoma (NHL), including any of the following subtypes:

  * Grade III follicular large cell lymphoma
  * Diffuse large B-cell lymphoma
  * Immunoblastic lymphoma
  * Plasmablastic lymphoma
  * Primary effusion lymphoma
* Previously untreated disease
* Any stage disease
* CD20 positive disease
* Must have documented HIV infection

  * Documentation may be by serology (enzyme-linked immunosorbent assay, western blot), culture, or quantitative polymerase chain reaction or branched DNA assays
  * Prior documentation of HIV seropositivity allowed
* Measurable or nonmeasurable disease
* Currently receiving effective highly active anti-retroviral therapy
* No primary CNS lymphoma, including parenchymal brain or spinal cord lymphoma
* No presence of leptomeningeal disease (positive cerebrospinal fluid for lymphoma) or presence of metastatic disease to brain, in terms of any mass lesion

PATIENT CHARACTERISTICS:

* ECOG performance status (PS) 0-2 OR Karnofsky PS 50-100%
* Life expectancy ≥ 2 months
* Absolute granulocyte (neutrophil) count ≥ 1,000/mm³ (unless secondary to lymphomatous involvement of bone marrow)
* Platelet count ≥ 75,000/mm³ (unless secondary to lymphomatous involvement of bone marrow or due to HIV-related thrombocytopenia)
* Bilirubin ≤ 2.0 mg/dL (unless elevated secondary to lymphomatous involvement of liver or biliary system or due to other HIV medications [e.g., indinavir, tenofavir, or atazanavir])
* SGOT ≤ 5 times upper limit of normal
* Creatinine ≤ 2.0 mg/dL OR creatinine clearance ≥ 60 mL/min (unless secondary to renal involvement by lymphoma)
* LVEF normal by MUGA or echocardiogram
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 6 months after completion of study treatment
* No other malignancy, except nonmelanoma skin cancer, carcinoma in situ of the cervix, or Kaposi's sarcoma that does not require systemic therapy
* No serious, ongoing, nonmalignant disease or infection that would preclude study compliance, in the opinion of the investigator
* No history of cutaneous or mucocutaneous reactions, or diseases in the past, due to any cause, severe enough to cause hospitalization or an inability to eat or drink for ≥ 2 days
* No acute, intercurrent infection that would preclude study treatment

  * Patients with Mycobacterium avium are eligible
* No cardiovascular problems, including any of the following:

  * Myocardial infarction within the past 6 months
  * New York Heart Association class II-IV heart failure
  * Uncontrolled angina
  * Severe uncontrolled ventricular arrhythmias
  * Clinically significant pericardial disease
  * ECG evidence of acute ischemic or active conduction system abnormalities.
* No shortness of breath at rest
* Arterial PO_2 ≥ 70 or pulse oximeter-derived O_2 saturation ≥ 94% on room air (unless due to lymphomatous involvement of the lungs)
* Able to comply with study and provide adequate informed consent

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* At least 4 weeks since prior major surgery (except diagnostic surgery)
* At least 12 months since prior rituximab unless it was only given for indications other than the treatment of aggressive lymphoma
* No prior cytotoxic chemotherapy or radiotherapy for this lymphoma

  * Concurrent radiotherapy, with or without steroids, for emergency conditions secondary to lymphoma (i.e., CNS tumor or cord compression) allowed
* No zidovudine or zidovudine-containing regimen (including Combivir® or Trizivir®) during and for 2 months after completion of chemotherapy
* Concurrent erythropoietin or filgrastim (G-CSF) allowed

  * Growth factor therapy must be discontinued ≥ 24 hours prior to study entry

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2007-01; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra M. Levine, MD, Study Chair — City of Hope Comprehensive Cancer Center
Locations (14):
- United States (14):
  - Rebecca and John Moores UCSD Cancer Center, La Jolla, California
  - USC/Norris Comprehensive Cancer Center and Hospital, Los Angeles, California
  - UCLA Clinical AIDS Research and Education (CARE) Center, Los Angeles, California
  - University of Miami Sylvester Comprehensive Cancer Center - Miami, Miami, Florida
  - Robert H. Lurie Comprehensive Cancer Center at Northwestern University, Chicago, Illinois
  - Ochsner Cancer Institute at Ochsner Clinic Foundation, New Orleans, Louisiana
  - Boston University Cancer Research Center, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Siteman Cancer Center at Barnes-Jewish Hospital - Saint Louis, St Louis, Missouri
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Albert Einstein Cancer Center at Albert Einstein College of Medicine, The Bronx, New York
  - Case Comprehensive Cancer Center, Cleveland, Ohio
  - Joan Karnell Cancer Center at Pennsylvania Hospital, Philadelphia, Pennsylvania
  - Virginia Mason Medical Center, Seattle, Washington

REFERENCES:
- [Result] Levine AM, Noy A, Lee JY, Tam W, Ramos JC, Henry DH, Parekh S, Reid EG, Mitsuyasu R, Cooley T, Dezube BJ, Ratner L, Cesarman E, Tulpule A. Pegylated liposomal doxorubicin, rituximab, cyclophosphamide, vincristine, and prednisone in AIDS-related lymphoma: AIDS Malignancy Consortium Study 047. J Clin Oncol. 2013 Jan 1;31(1):58-64. doi: 10.1200/JCO.2012.42.4648. Epub 2012 Nov 19. PMID 23169503

RESULTS

PARTICIPANT FLOW:
Groups:
- DR-COP: Single arm interventional study: all subjects receive Doxil, Rituximab, Cyclophosphamide, Vincristine and Prednisone (DR-COP) regimen.
Period: Overall Study
Arm/Group | DR-COP
Started | 43
Completed | 40
Not Completed | 3

BASELINE CHARACTERISTICS:
Arm/Group | DR-COP
Number analyzed (Participants) | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 39
  >=65 years | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.4 (8.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 30
Region of Enrollment [Number; unit: participants]
  United States | 40

OUTCOME MEASURES:

1. Primary Outcome: Complete Response Rate (Complete Response and Complete Response Unconfirmed) Defined as Disappearance of All Evidence of Disease Based on Radiographic Findings on CT or MRI .
Time Frame: After cycles 2, 4, 6, 1 month after treatment discontinuation, every 2 months for 1 year after treatment discontinuation, every 6 months during the second and third years after treatment discontinuation
Measure: Number (95% Confidence Interval); unit: proportion of patients
Arm/Group | DR-COP
Number analyzed (Participants) | 40
proportion of patients | 0.475 [0.315 to 0.639]

2. Primary Outcome: Duration of Response
Time Frame: as for outcome 1
Reporting Status: Not Posted

3. Primary Outcome: Median Survival Time
Time Frame: as for outcome 1
Reporting Status: Not Posted

4. Primary Outcome: Rate of Bacterial, Fungal, and Opportunistic Infections
Time Frame: After every cycle of treatment, 1 month after treatment discontinuation, every 2 months for 1 year after treatment discontinuation, every 6 months during the second and third years after treatment discontinuation
Reporting Status: Not Posted

5. Secondary Outcome: Relationship Between MDR-1 Expression and Response to Treatment
Time Frame: Baseline
Reporting Status: Not Posted

6. Secondary Outcome: Relationship Between Response and Survival and BCL-2 Expression in Tumor Tissue
Time Frame: Baseline, after cycles 4 and 6, 1 month after treatment discontinuation
Reporting Status: Not Posted

7. Secondary Outcome: Relationship Between Development of Bacterial, Fungal, and/or Opportunistic Infections and Baseline CD4 Lymphocyte Count, HIV-1 RNA Level, and Quantitative Immunoglobin Level, or Changes in Quantitative Immunoglobin Levels Over Time
Time Frame: as for outcome 4
Reporting Status: Not Posted

8. Secondary Outcome: Mortality and Cause of Death
Time Frame: At any time through the third year after treatment discontinuation
Reporting Status: Not Posted

9. Secondary Outcome: Event-free Survival at 1 Year
Time Frame: 1 year post-treatment
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | DR-COP
Serious Adverse Events (participants affected / at risk) | 26/40
Other Adverse Events (participants affected / at risk) | 38/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DR-COP (N=40)
Anemia (Blood and lymphatic system disorders) | 2 (2)
Febrile Neutropenia (Blood and lymphatic system disorders) | 3 (4)
Optic nerve disorder (Eye disorders) | 1 (3)
Abdominal pain (Gastrointestinal disorders) | 2 (3)
Constipation (Gastrointestinal disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Gastric hemorrhage (Gastrointestinal disorders) | 1 (1)
Ileal obstruction (Gastrointestinal disorders) | 1 (1)
Ileal perforation (Gastrointestinal disorders) | 1 (1)
Ileus (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (3)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 3 (5)
Death (General disorders) | 12 (12)
Fever (General disorders) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1)
Pain (General disorders) | 1 (1)
Abdominal infection (Infections and infestations) | 1 (1)
Cather related infection (Infections and infestations) | 2 (2)
Lung infection (Infections and infestations) | 1 (1)
Skin infection (Infections and infestations) | 1 (1)
Neutrophil count decreased (Investigations) | 6 (9)
Platelet count decreased (Investigations) | 3 (4)
Weight loss (Investigations) | 2 (3)
White blood cell decreased (Investigations) | 3 (3)
Dehydration (Metabolism and nutrition disorders) | 2 (2)
Hyperuricemia (Metabolism and nutrition disorders) | 1 (1)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (2)
Headache (Nervous system disorders) | 1 (1)
Intracranial hemorrhage (Nervous system disorders) | 1 (1)
Leukoencephalopathy (Nervous system disorders) | 1 (1)
Peripheral motor neuropathy (Nervous system disorders) | 2 (5)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1)
Seizure (Nervous system disorders) | 1 (1)
Confusion (Psychiatric disorders) | 1 (1)
Delirium (Nervous system disorders) | 1 (1)
Cystitis noninfective (Renal and urinary disorders) | 1 (1)
Renal and urinary disorders, other (Renal and urinary disorders) | 1 (1)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4 (6)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DR-COP (N=40)
Anemia (Blood and lymphatic system disorders) | 13 (19)
Abdominal pain (Gastrointestinal disorders) | 5 (6)
Nausea (Gastrointestinal disorders) | 13 (19)
Vomiting (Gastrointestinal disorders) | 12 (17)
Blood and lymphatic system disorders, other (Blood and lymphatic system disorders) | 3 (6)
Sinus tachycardia (Cardiac disorders) | 2 (2)
Ear and labyrinth disorders, other (Ear and labyrinth disorders) | 2 (2)
Constipation (Gastrointestinal disorders) | 11 (14)
Diarrhea (Gastrointestinal disorders) | 7 (8)
Dysphagia (Gastrointestinal disorders) | 3 (3)
Gastric ulcer (Gastrointestinal disorders) | 2 (2)
Mucositis, oral (Gastrointestinal disorders) | 6 (10)
Chills (General disorders) | 6 (6)
Edema, limbs (General disorders) | 5 (6)
Fatigue (General disorders) | 14 (19)
Fever (General disorders) | 8 (10)
Non-cardiac chest pain (General disorders) | 2 (2)
Pain (General disorders) | 3 (4)
Infections and investigations, other (Infections and infestations) | 4 (4)
Mucosal infections (Infections and infestations) | 5 (5)
Upper respiratory infection (Infections and infestations) | 2 (2)
Urinary tract infection (Infections and infestations) | 2 (2)
Alanine aminotransferase increased (Investigations) | 3 (4)
Alkaline phosphatase increased (Investigations) | 3 (3)
Aspartate aminotransferase increased (Investigations) | 3 (3)
Lymphocyte count decreased (Investigations) | 6 (18)
Neutrophil count decreased (Investigations) | 22 (54)
Platelet count decreased (Investigations) | 3 (4)
Weight gain (Investigations) | 2 (3)
Weight loss (Investigations) | 7 (10)
White blood cell decreased (Investigations) | 10 (30)
Anorexia (Metabolism and nutrition disorders) | 6 (8)
Dehydration (Metabolism and nutrition disorders) | 3 (3)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (3)
Bone pain (Musculoskeletal and connective tissue disorders) | 3 (4)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 (6)
Headache (Nervous system disorders) | 8 (13)
Leukoencephalopathy (Nervous system disorders) | 2 (2)
Memory impairment (Nervous system disorders) | 2 (2)
Peripheral motor neuropathy (Nervous system disorders) | 3 (4)
Peripheral sensory neuropathy (Nervous system disorders) | 13 (19)
Anxiety (Psychiatric disorders) | 3 (3)
Depression (Psychiatric disorders) | 2 (3)
Insomnia (Psychiatric disorders) | 5 (5)
Urinary frequency (Renal and urinary disorders) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 7 (8)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (5)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 5 (6)
Alopecia (Skin and subcutaneous tissue disorders) | 5 (5)
Dry skin (Skin and subcutaneous tissue disorders) | 4 (4)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 (3)
Nail loss (Skin and subcutaneous tissue disorders) | 2 (2)
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 5 (10)
Pruritus (Skin and subcutaneous tissue disorders) | 4 (4)
Skin and subcutaneous tissue disorders, other (Skin and subcutaneous tissue disorders) | 4 (5)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2011-01-21): https://cdn.clinicaltrials.gov/large-docs/18/NCT00389818/Prot_SAP_001.pdf